CLINICAL TRIAL: NCT06229769
Title: A Monocentric, Prospective, Longitudinal and Observational Natural History Study for Patients With Angelman Syndrome in CHR Citadelle Liège : NatHis-Angelman
Brief Title: Natural History Study for Patients With Angelman Syndrome
Acronym: NatHisAngelman
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Collaborators: Centre Hospitalier Régional de la Citadelle (Other); SYSNAV (Industry)
Responsible Party: Principal Investigator, Laurent Servais, Prof. Investigator of CRMN Liège, Principal investigator, Centre Hospitalier Universitaire de Liege
Other Study IDs: NatHis-Angelman
Record Dates: First submitted 2023-11-02; First posted 2024-01-29 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Angelman Syndrome
Keywords: Actimyo°; Accelerometry; Daily living
MeSH Terms: conditions — Angelman Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — One EDTA sample of 5ml at baseline visit only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study is a 9-year natural history study for patients with Angelman syndrome in Belgium (a genetic neurodevelopmental disorder, affecting 500,000 individuals in the world). It includes a 3-year recruitment phase, a 5 year follow-up and a year to analyze the collected data. The investigators plan to include 30 patients with a semi-annual follow-up for 4 years.

The investigators will collect relevant retrospective and prospective data using age-standardized scales and questionnaires for functional motor assessments and global developmental assessment.

DETAILED DESCRIPTION:
Patients are seen every six months for five years. In these visits, patient have medical review (general medical examination, neurological examination), vital signs (height, weight, respiratory rate, heart rate, blood pressure), cognitive assessment (Bayley-IV), language assessment and questionaire (Bayley-IV, ORCA), motor assessments (Bayley-IV, FMS, Developmental milestones and HINE), quality of life questionnaire (PedsQL, CGI-CASS) and general development questionnaire (Vineland-II).

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed diagnosis of AS
* 0-99 years
* Male or Female
* Participant's carer is willing to give IC/sign a "record of consultation" for participation in the study

Exclusion Criteria:

* comorbidity that could potentially affect the results of the study coexists. This

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Angelman Syndrom
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-10-10 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Bayley-IV gross motor functions | 2 years
  Scale of 58 items of Gross motor (raw score 0 to 116) development evaluation.
Bayley-IV fine motor functions | 2 years
  Scale of 46 items of fine motor scale (raw score 0 to 92) development evaluation.
Bayley-IV Cognitive | 2 years
  Scale of 81 items of cognitive scale development evaluation (raw score 0 to 162).
Bayley-IV Receptive Communication | 2 years
  Scale of 42 items of receptive communication abilities scale in development evaluation (raw score 0 to 84).
Bayley-IV Expressive Communication | 2 years
  Scale of 37 items of expressive communication abilities scale in development evaluation (raw score 0 to 74).
Functional Mobility Scale (FMS) | 2 years
  Scale o 3 items (5, 50 and 500 meters distance of ability to move alone) to classify children's functional mobility, document change over time in the same child and to document change seen following. This scale is scored 1 (moving alone with wheelchair) to 6 (running).
Developmental Milestones | 2 years
  Scale to Evaluate the general gross motor milestones of 6 items global motor ability, from ability to sit without support to walk alone (score by able or not able). .
Hammersmith Infant Neurological Examination (HINE - if under 2 years old) | 2 years
  Scale of 8 items to evaluation the mobility in young children, scored 0 (unable) to 4 (able and normal for children age) per items (total raw score from 0 to 32).
Vineland-II | 2 years
  11 subscales of items evaluated with Caregivers interview tool for assessing the level of autonomy and adaptation for all ages.
  Subscales are composed as following (higher scores with better the abilites):
  1. Listening and understanding, raw score 0 to 40;
  2. Speaking, raw score 0 to 108,
  3. Reading and writing, raw score 0 to 54,
  4. Self caring, raw score 0 to 82,
  5. Home caring, raw score 0 to 48,
  6. Community living, raw score 0 to 88,
  7. Contact with others, raw score 0 to 76,
  8. Play and use your free time, raw score 0 to 62,
  9. Adapting, raw score 0 to 60,
  10. Gros motor, raw score 0 to 80,
  11. Fine motor, raw score 0 to 72,
Observed Reported Communication Assessment (ORCA) | 2 years
  Caregivers interview of 23 items with subscales to assessing the general communication.
  This is a qualitative questionnaire.
Continuous movement monitoring using ActiMyo® | 2 years
  To improve the design of future clinical trials by validating tools of assessment based on their suitability to be used as prognostic measures.

SECONDARY OUTCOMES:
Clinical Global Impression - Improvement - Angelman Syndrome (CGI-I-AS) | 2 years
  Caregivers interview of quality of life severity and change in patient with Angelman Syndrome since last 7 days and since the last month.
  Part regarding the severity in last 7 days is composed of 9 items scored 0 ("not at all difficult") to 4 ("very difficult"), raw score is between 0 to 36.
  Part regarding change in last month is composed of 9 items scored 1 ("very much improved") to 7 ("very much worse"), raw score is between 0 to 63,
Pediatric Quality of Life (PedsQL) | 2 years
  Caregivers interview of quality of life and family impact in daily life separated in two parts, one regarding the last 7 days and one regarding the last month.
  Total raw score for each part is on 100 (100 related to no impact to 0 related to a huge impact).

OTHER OUTCOMES:
Blood sample collection and DNA extraction and storage | 1 year
  To create a DNA biobank

CONTACTS AND LOCATIONS:
Overall Officials: Laura Vanden Brande, Principal Investigator — CHR Citadelle
Locations (1):
- CHR Citadelle Liège, Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No